CLINICAL TRIAL: NCT07310888
Title: Robotic Gastrectomy With a Novel 5th Arm - an International Multicenter Pilot Study
Brief Title: Robotic Gastrectomy With 5th Arm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2025.666
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5th arm group (Experimental)
  Interventions: Device: Robotic gastrectomy performed with Cornerstone Robotics Sentire Surgical System C1000 Ultra (With Patient Side Single Arm)

INTERVENTIONS:
Device: Robotic gastrectomy performed with Cornerstone Robotics Sentire Surgical System C1000 Ultra (With Patient Side Single Arm) — Under general anesthesia, the patient will be placed in a supine position in reverse Trendelenburg tilt. A 25-mm transumbilical incision will be made to allow placement of a GelPOINT Mini Advanced Access Platform (Applied Medical Ltd) and introduction of capno-peritoneum. Through the GelPOINT seal cap, robotic 8-10mm camera port and an accessory 12mm port will be introduced. Laparoscopic insertion of the other four ports of 8 mm for placement of robotic arms will be performed. After confirming port positions, docking of the Sentire Surgical System C1000 Ultra would be performed. The main Patient Side Robot (PSR) will be introduced from the patient's left shoulder side, while the Patient Side Single Arm will be introduced from the patient's right side. Distal gastrectomy, total gastrectomy and proximal gastrectomy will be performed according to the Japanese Treatment Guidelines of Gastric Cancer.

SUMMARY:
This is a multicenter single arm clinical pilot study to investigate the safety and feasibility of a novel multiport Sentire Robotic Surgical System with Patient Side Single Arm (5th arm) in patients with gastric cancer undergoing robotic radical gastrectomy. 10 adult patients with newly diagnosed cancer of the stomach deemed operable would be recruited from Prince of Wales Hospital, Hong Kong and Fujita Health University Hospital, Nagoya, Japan.

The primary aim of this study is to determine the feasibility of robotic surgical procedures performed using the Cornerstone Robotics Sentire Surgical System C1000 Ultra, as measured by the technical success rate of surgery, and to evaluate the safety of the procedures as measured by the incidence of perioperative complications.

DETAILED DESCRIPTION:
Laparoscopic surgery is a well-established minimally invasive surgery (MIS) technique, and is currently the standard treatment approaches for various benign and malignant surgical diseases of the abdomen [1]. In comparison with traditional open surgery, where a large surgical incision is made, laparoscopic surgery uses three to six small (0.5-1.5 cm) incisions to complete similar operative procedures. Based on numerous randomized controlled trials, minimally invasive surgeries have been proven to be beneficial in reducing patient trauma and morbidity, expediting postoperative recovery, and improving cosmesis when compared with open surgery [2,3].

The quest to develop precise and safe MIS in order to further reduce surgical trauma and improve patients' outcome still remains robust. Robotic technologies are expected to overcome the technical challenges associated with conventional laparoscopic surgery, including the limitation in degree of freedom associated with conventional laparoscopic instruments as well as lack of precision for dissection. The da Vinci Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA, USA) was initially developed in 1999 to address the technical disadvantages of conventional laparoscopic surgery in terms of visualization and maneuverability. The robotic system provides a stable camera platform with magnified 3D view, and intuitively transfers movements from the handle to the tip of the instrument with tremor filtering. Dexterity is enhanced via EndoWrist technology, returning seven degrees of freedom to the surgeon [4].

Despite its technical advantages, robotic surgery has always been criticized for being highly expensive, which has limited its accessibility and wider applications [5,6]. The current da Vinci Surgical System from Intuitive Surgical has high performance with excellent quality. However, the high cost for each robotic surgical procedure has imposed major financial impact to patients and hospitals. In order to provide a cost-effective solution, introduction of new robotic systems with similar quality of performance and lower instalment /maintenance costs is necessary.

Robotic Surgery in Gastric Cancer Surgery Laparoscopic surgery, is widely accepted as curative treatment for gastric cancer (GC). Several multicentre randomized clinical trials (RCTs) have reported lower rates of postoperative complications in patients who underwent laparoscopic gastrectomy (LG) compared with open gastrectomy, but with similar long-term prognosis between them [7-11]. Laparoscopic gastrectomy still has several drawbacks, however, including the limited range of movement, amplification of operator hand tremors, and inconvenient surgical positioning [12-16]. Specifically, for D2 lymphadenectomy, laparoscopic instruments lack the dexterity during supra-pancreatic dissection leading to pancreatic injury [12-13].

With the technical advantages described above, robotic gastrectomy (RG) may therefore overcome some of the drawbacks associated with LG. An RCT from China has shown that RG is associated with better short term outcomes such as lower morbidity rate, faster recovery, milder inflammatory responses, and improved lymphadenectomy [17]. The 3-year oncological outcome of the same trial also showed that RG has improved 3-year DFS and cumulative recurrence rate [18]. Another RCT from Japan reported a significantly lower postoperative surgical complications of Clavien-Dindo Grade II or higher although did not show difference in intra-abdominal infectious complications [19].

Sentire Surgical System

The Cornerstone Robotics Sentire Surgical System [C1000], developed by Cornerstone Robotics Limited (https://www.csrbtx.com), is a software-controlled, electro-mechanical system designed for surgeons to perform minimally invasive surgery in the thorax and abdomen. It consists of 1 or 2 Surgeon Console(s) [SGC], a Patient Side Robot [PSR], and a Vision Cart [VCT], and is intended for use with an endoscope, Surgical Instruments [SGI], and Accessories [ACC]. Surgeons view the 3D endoscopic image through a High-resolution Stereo Viewer, which provides a view of the abdominal/thoracic cavity and surgical instrumentation, enhanced by icons and various user interface features that facilitate navigation and control.

The VCT contains electronic and video processing equipment, while the PSR is positioned at the operating room, featuring four arms equipped with instrument drives for attaching surgical instruments or the endoscope. The PSR is then positioned over the target patient anatomy. The endoscope provides the surgeon with a high-resolution 3D view. A suite of surgical instruments can be easily attached to and detached from the other three arms, enabling surgeons to perform various surgical tasks. The endoscope and up to three instruments can be used simultaneously, entering the patient through separate 8-mm or 10-mm cannulae.

The surgical instruments come in configurations such as graspers, scissors, and needle drivers, featuring an unique articulating design at the distal tip that mimics the human wrist, shoulder, and elbow for triangulation and X-Y-Z movement. Each instrument is designated for specific surgical tasks, such as grasping, suturing, tissue manipulation, and electrosurgery. They are reusable and designed exclusively for the Sentire Surgical System, programmed for a maximum number of procedures based on life testing. The endoscope is reusable, and it provides a stereo image of the surgical site.

After completion of pre-clinical and prospective clinical trials using the Sentire Surgical System (C1000) in Hong Kong (By the CUHK Team), and mainland China based on the Innovation, Development, Exploration, Assessment, Long-term Study (IDEAL) Collaboration group methodology, Cornerstone Robotics Limited obtained National Medical Products Administration (NMPA) approval in China for Sentire Surgical System C1000 in September 2024.

Concept of 5th arm (Patient Side Single Arm)

The Patient Side Single Arm [PSR-SA] is an independent robotic arm designed for compatibility with the C1000, creating the hybrid surgical system known as the C1000 Ultra. With 14 degrees of freedom (DoF) and a software remote center design, it enhances port placement flexibility, minimizes arm collisions with the patient or operating table, and optimizes docking for seamless integration into the operating room.

The PSR-SA provides full compatibility with a range of surgical instruments, including graspers, scissors, needle drivers, and endoscopes, ensuring versatility in surgical procedures. Control of the hybrid system can be managed from either a single console or a dual console setup, depending on the surgeon's preference. The 4+1 configuration empowers surgeons by effectively acting as a "fifth robotic arm," enabling them to realize new surgical and bedside possibilities directly from the console.

The dual console configuration facilitates collaboration between two surgeons, enabling simultaneous control of all robotic arms with a shared high-resolution 3D view of the surgical site. It in turn allows both surgeons to align their angles of approach, significantly enhancing coordination and precision during procedures. By fostering teamwork and communication, this innovative system improves the effectiveness of complex surgeries, ultimately leading to better patient outcomes.

Pre-clinical Data on Cornerstone Robotics Sentire Surgical System [C1000 Ultra]

Preclinical studies, including cadaveric model studies, have been completed by our team of surgeons from the Department of Surgery, Faculty of Medicine, The Chinese University of Hong Kong. Between March and July 2025, nine robotic procedures in colorectal surgery, urology, hepatobiliary, and upper gastrointestinal surgery were performed using cadaveric models, at the Multi-scale Medical Robotics Center in the Hong Kong Science & Technology Park. In particular, two robotic gastrectomies and one robotic esophagectomy was completed using the system.

The studies evaluated the safety and efficacy of C1000 Ultra, with which the surgeons successfully completed all procedures. Clinical feedback on the system's performance was collected using a Likert-scale questionnaire, with scores ranging from 1 to 5. The acceptance criterion was a score higher than 3, with higher scores indicating more positive feedback. The mean scores across nine domains - surgical instruments, control, hardware usability, compatibility with standard operational infrastructure, hardware performance, safety, software user interface, vision, and overall satisfaction - met the acceptance criteria.

Based on the encouraging results from pre-clinical studies using the Sentire Surgical System C1000 Ultra, the investigators plan to conduct the first multi-center clinical trial using the system for radical gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Body mass index <35 kg/m2
* Newly diagnosed tumors of the stomach / gastro-esophageal junction, scheduled to undergo elective gastrectomy (Proximal gastrectomy, distal gastrectomy, total gastrectomy)
* Willingness to participate as demonstrated by giving informed consent

Exclusion Criteria:

* Previous abdominal surgery precluding performance of MIS gastrectomy
* Contraindication to general anesthesia
* Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
* Untreated active infection
* Noncorrectable coagulopathy
* Presence of another malignancy or distant metastasis
* Emergency surgery
* Vulnerable population (e.g., mentally disabled, pregnancy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Technical success | 1 day
  Successful completion of the intended surgical procedure using the Sentire Surgical System C1000 Ultra, without conversion the treatment plan to conventional minimally invasive laparoscopic surgery or to open surgery.

SECONDARY OUTCOMES:
Intra-operative complication | 1 day
  The rate of intra-operative complications
Post-procedural complication | 30 days or in-hospital
  The rate of post-procedural complication, as graded by Clavien Dindo Classification
Operative time | 1 day
  Procedure time of the robotic gastrectomy
Intraoperative blood loss | 1 day
  The volume of blood loss estimated during procedure (ml)
Post-operative pain score | 7 days
  Postoperative pain evaluated on a Visual Analogue scale
Post-procedure hospital stay | 3 months
  Duration of hospital stay after the procedure (Days)
Resection margin status | 30 days
  The clearance of resection margin on histology
Lymph node harvest | 30 days
  The total number of lymph node harvested from pathology
Cancer Recurrence | 2 years
  The recurrence of cancer detected on postoperative CT scan or by histology.

CONTACTS AND LOCATIONS:
Locations (2):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Fujita Health University Hospital, Nagoya, Japan

IPD SHARING:
Plan to Share IPD: No